CLINICAL TRIAL: NCT00935818
Title: Combination Therapy With Varenicline and Bupropion for Smoking Cessation
Brief Title: Varenicline and Bupropion for Smoking Cessation
Acronym: CHANBAN
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH); University of Minnesota (Other)
Responsible Party: Principal Investigator, Jon Ebbert, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 09-003598; 09-002459 (Other: Mayo Clinic IRB number); 1R01CA138417 (NIH)
Record Dates: First submitted 2009-07-06; First posted 2009-07-09 (Estimated); Results first posted 2014-04-24 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2014-04

CONDITIONS: Smoking
Keywords: smoking; nicotine; tobacco; dependence; cessation; abstinence
MeSH Terms: conditions — Smoking | interventions — Varenicline; Sugars; Bupropion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- varenicline and buproprion SR (Active Comparator): Everyone randomized to this arm will receive varenicline (up to 1mg bid) and bupropion SR (150 mg bid)for 12 weeks. They will be followed up by study for an additional 9 months post end of medication - for a total of 1 year study participation. Everyone will receive behavioral counseling for the full year.
  Interventions: Drug: Varenicline; Drug: bupropion SR
- varenicline and placebo (Placebo Comparator): Everyone randomized to this arm will receive varenicline (up to 1mg bid) and placebo (0 mg bid)for 12 weeks. They will be followed up by study for an additional 9 months post end of medication - for a total of 1 year study participation. Everyone will receive behavioral counseling for the full year.
  Interventions: Drug: Varenicline; Drug: placebo

INTERVENTIONS:
Drug: Varenicline — varenicline - 1 mg bid for 12 weeks
  Other Names: chantix
Drug: placebo — placebo for 12 weeks
  Other Names: sugar pill
  Arms: varenicline and placebo
Drug: bupropion SR — bupropion sr - 150 mg bid for 12 weeks
  Other Names: wellbutrin SR; zyban
  Arms: varenicline and buproprion SR

SUMMARY:
This study provides an opportunity to combine varenicline and bupropion SR and capitalize on the potential additive benefit. The investigators hypothesize that this will further increase long-term (≥ 6 months) smoking abstinence rates.

DETAILED DESCRIPTION:
Cigarette smoking is the single most important preventable cause of morbidity, mortality and excess health care costs in the United States and accounts for 30% of U.S. cancer deaths. Varenicline and bupropion SR (sustained-release) are non nicotine pharmacotherapies FDA-indicated for the treatment of tobacco dependence in cigarette smokers. Although varenicline has proven greater efficacy than bupropion SR, both medications are associated with high end-of-treatment smoking abstinence rates. However, almost two-thirds of smokers treated with varenicline report smoking at 6 months. Because varenicline and bupropion SR have different mechanisms of action and different neuropharmacologic targets, combination pharmacotherapy with these agents may increase long-term smoking abstinence rates above what is observed with single-agent therapy. In our recent pilot study of combination therapy with varenicline and bupropion SR, we observed treatment to be well-tolerated with 7-day point prevalence smoking abstinence rates of 71% (95% CI: 54-85%) at 3 months and 58% (95% CI: 41-74%) at 6 months. Determining the efficacy of combination therapy compared to single-agent therapy has immediate and important clinical implications. In this study, we will conduct a randomized, multicenter, controlled clinical trial evaluating the efficacy of combination therapy with varenicline and bupropion SR compared to varenicline and placebo in 506 cigarette smokers at the Mayo Clinic in Rochester, MN, and the University of Minnesota in Minneapolis, MN.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is at least 18 years of age;
2. Subject has provide written informed consent;
3. Subject is smoking greater than or equal to 10 cigarettes per day for at least 6 months;

3) Subject is able to complete all study visits 4) Subject is in good health as determined by the investigator 5) Subject has the ability to participate fully in all aspects of the study and keep scheduled appointments 6) Subject is motivated to stop smoking.

Exclusion Criteria:

Female and were pregnant, lactating or likely to become pregnant during the trial and not able nor willing to use contraception or had:

1. an unstable medical condition;
2. another household member participating in the study;
3. bupropion or varenicline allergy;
4. current use (previous 30 days) of a tobacco dependence treatment and unable or unwilling to discontinue use;
5. an unstable medical condition or unstable angina, myocardial infarction, or coronary angioplasty (past 3 months) or an untreated cardiac dysrhythmia;
6. a history of renal failure or were on renal dialysis;
7. a history of seizures;
8. as defined by the C-SSRS (Columbia-Suicide Severity Rating Scale), current non-specific suicidal thoughts or lifetime history of a suicidal attempt (defined as "potentially self-injurious act committed with at least some wish to die, as a result of act");
9. a history of closed head trauma associated with > 30 minutes of loss of consciousness, amnesia, skull fracture, subdural hematoma, or brain contusion;
10. a history or psychosis, bipolar disorder, bulimia or anorexia nervosa;
11. current moderate or severe depression as assessed by a score of ≥ 20 on the Beck Depression Inventory, Second Edition (BDI-II) 10;
12. active substance abuse other than nicotine;
13. current (past 14 days) use of an antipsychotic, monoamine oxidase inhibitors, or drugs known to interact with bupropion SR;
14. a recent dose change of their antidepressant (within last 3 months);
15. untreated hypertension or baseline systolic blood pressure > 180 or diastolic > 100;
16. current treatment with another investigational drug for tobacco dependence (previous 30 days); or
17. current use of bupropion or varenicline (previous 30 days).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 506 (Actual)
Dates: Start 2009-09; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jon Ebbet, MD, Principal Investigator — Mayo Clinic; Dorothy Hatsukami, PhD, Study Director — University of Minnesota
Locations (3):
- United States (3):
  - University Of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Franciscan Skemp Hospital, La Crosse, Wisconsin

REFERENCES:
- [Result] Ebbert JO, Hatsukami DK, Croghan IT, Schroeder DR, Allen SS, Hays JT, Hurt RD. Combination varenicline and bupropion SR for tobacco-dependence treatment in cigarette smokers: a randomized trial. JAMA. 2014 Jan 8;311(2):155-63. doi: 10.1001/jama.2013.283185. PMID 24399554
- [Derived] Livingstone-Banks J, Fanshawe TR, Thomas KH, Theodoulou A, Hajizadeh A, Hartman L, Lindson N. Nicotine receptor partial agonists for smoking cessation. Cochrane Database Syst Rev. 2023 May 5;5(5):CD006103. doi: 10.1002/14651858.CD006103.pub8. PMID 37142273
- [Derived] Hartmann-Boyce J, Theodoulou A, Farley A, Hajek P, Lycett D, Jones LL, Kudlek L, Heath L, Hajizadeh A, Schenkels M, Aveyard P. Interventions for preventing weight gain after smoking cessation. Cochrane Database Syst Rev. 2021 Oct 6;10(10):CD006219. doi: 10.1002/14651858.CD006219.pub4. PMID 34611902

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was between October 2009 and April 2012. Volunteers from local communities of Rochester, MN, Minneapolis, MN and LaCrosse, WI, were recruited using newspaper classified ads, radio, TV, internet ads, print ads in magazines, word of mouth, and volunteer wait lists.
Pre-assignment Details: Study subjects who consented, were screened for entry criteria, and asked to return for a physical exam and medical history. If eligible and still interested, the volunteer was asked to return to the baseline visit at which time they would receive the study medication assignment.
Groups:
- Varenicline and Buproprion SR: Everyone randomized to this arm will receive varenicline (up to 1mg bid) and bupropion SR (150 mg bid)for 12 weeks. They will be followed up by study for an additional 9 months post end of medication - for a total of 1 year study participation. Everyone will receive behavioral counseling for the full year.
  varenicline and bupropion: varenicline - 1 mg bid for 12 weeks bupropion sr - 150 mg bid for 12 weeks
- Varenicline and Placebo: Everyone randomized to this arm will receive varenicline (up to 1mg bid) and placebo (0 mg bid)for 12 weeks. They will be followed up by study for an additional 9 months post end of medication - for a total of 1 year study participation. Everyone will receive behavioral counseling for the full year.
  varenicline and placebo: varenicline (1 mg bid) for 12 weeks placebo for 12 weeks
Period: Overall Study
Arm/Group | Varenicline and Buproprion SR | Varenicline and Placebo
Started | 249 | 257
End of Medication Phase | 182 | 184
Completed | 158 | 157
Not Completed | 91 | 100
Not completed — Withdrawal by Subject | 45 | 50
Not completed — Lost to Follow-up | 40 | 42
Not completed — Adverse Event | 6 | 7
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Population: Smokers from the local community who smoked 10 cigarettes or more per day for the 6 months prior to study entry.
Groups:
- Total: Total of all reporting groups
Arm/Group | Varenicline and Buproprion SR | Varenicline and Placebo | Total
Number analyzed (Participants) | 249 | 257 | 506
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 0 | 3
  Between 18 and 65 years | 234 | 253 | 487
  >=65 years | 12 | 4 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.2 (12.2) | 41.9 (12.7) | 42.1 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 113 | 126 | 239
  Male | 136 | 131 | 267
Race/Ethnicity, Customized [Number; unit: participants]
  White, non-hispanic | 234 | 240 | 474
  other | 15 | 17 | 32
smoking rate [Mean (Standard Deviation); unit: cigarettes per day] | 19.5 (7.3) | 19.7 (7.9) | 19.6 (7.6)

OUTCOME MEASURES:

1. Primary Outcome: Prolonged Smoking Abstinence Rates at 12 Weeks in Cigarettes Smokers.
Description: Prolonged smoking abstinence is defined as no smoking, not even a puff, in the last 7 days, and a negative response to the question "Since 2 weeks after your target quit date, have you smoked any tobacco, even a puff, for 7 consecutive days or at least once each week on 2 consecutive weeks?"
Time Frame: 3 months
Population: intention-to-treat (all randomized subjects included)
Measure: Number; unit: participants
Arm/Group | Varenicline and Buproprion SR | Varenicline and Placebo
Number analyzed (Participants) | 249 | 257
participants | 132 | 111
Statistical Analysis 1: Comparison: Varenicline and Buproprion SR vs Varenicline and Placebo; Logistic regression with covariate included for study site; Test type: Superiority or Other; p = 0.03, Regression, Logistic; Odds Ratio (OR) = 1.49, 95% CI 2-sided [1.05 to 2.12]

2. Secondary Outcome: Prolonged Smoking Abstinence Rates at 26 Weeks in Cigarettes Smokers.
Time Frame: 6 months
Population: intention to treat - all subjects
Measure: Number; unit: participants
Arm/Group | Varenicline and Buproprion SR | Varenicline and Placebo
Number analyzed (Participants) | 249 | 257
participants | 91 | 71
Statistical Analysis 1: Comparison: Varenicline and Buproprion SR vs Varenicline and Placebo; Logistic Regression - adjusting for study site; Test type: Superiority or Other; p = 0.03, Regression, Logistic; Odds Ratio (OR) = 1.52, 95% CI 2-sided [1.04 to 2.22]

3. Secondary Outcome: Weight Gain From Baseline to 3 Months
Description: Weight change from baseline to three months in those who met criteria for prolonged abstinence at the 3 month visit
Time Frame: 3 months
Population: analysis was restricted to subjects who had weight measured at the 3 month visit and were classified as meeting criteria for prolonged abstinence
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Varenicline and Buproprion SR | Varenicline and Placebo
Number analyzed (Participants) | 131 | 111
kilograms | 1.1 (3.4) | 2.5 (2.7)
Statistical Analysis 1: Comparison: Varenicline and Buproprion SR vs Varenicline and Placebo; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

4. Primary Outcome: Point Prevalence Abstinence at 3 Months.
Description: biochemically confirmed 7-day point prevalence abstinence defined as no smoking, not even a puff, in the previous 7 days.
Time Frame: 3 months
Population: intent to treat - all subjects
Measure: Number; unit: participants
Arm/Group | Varenicline and Buproprion SR | Varenicline and Placebo
Number analyzed (Participants) | 249 | 257
participants | 140 | 125
Statistical Analysis 1: Comparison: Varenicline and Buproprion SR vs Varenicline and Placebo; Logistic regression adjusted for study site; Test type: Superiority or Other; p = 0.09, Regression, Logistic; Odds Ratio (OR) = 1.36, 95% CI 2-sided [0.95 to 1.93]

5. Secondary Outcome: Point Prevalence Abstinence at 6 Months.
Description: Biochemically confirmed abstinence as no smoking, even a puff, for the prior 7 days.
Time Frame: 6 months
Population: Intention to treat - all subjects
Measure: Number; unit: participants
Arm/Group | Varenicline and Buproprion SR | Varenicline and Placebo
Number analyzed (Participants) | 249 | 257
participants | 95 | 82
Statistical Analysis 1: Comparison: Varenicline and Buproprion SR vs Varenicline and Placebo; Logistic Regression adjusting for study site; Test type: Superiority or Other; p = 0.14, Regression, Logistic; Odds Ratio (OR) = 1.32, 95% CI 2-sided [0.91 to 1.91]

6. Secondary Outcome: Prolonged Abstinence at 12 Months
Time Frame: 12 months
Population: intention to treat - all subjects
Measure: Number; unit: participants
Arm/Group | Varenicline and Buproprion SR | Varenicline and Placebo
Number analyzed (Participants) | 249 | 257
participants | 77 | 63
Statistical Analysis 1: Comparison: Varenicline and Buproprion SR vs Varenicline and Placebo; Logistic Regression - adjusting for study site; Test type: Superiority or Other; p = 0.11, Regression, Logistic; Odds Ratio (OR) = 1.39, 95% CI 2-sided [0.93 to 2.07]

7. Secondary Outcome: Point Prevalence Abstinence at 12 Months
Description: Biochemically confirmed abstinence defined as no smoking, not even a puff, in the last 7 days
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | Varenicline and Buproprion SR | Varenicline and Placebo
Number analyzed (Participants) | 249 | 257
participants | 91 | 75
Statistical Analysis 1: Comparison: Varenicline and Buproprion SR vs Varenicline and Placebo; Logistic Regression - adjusting for site; Test type: Superiority or Other; p = 0.08, Regression, Logistic; Odds Ratio (OR) = 1.40, 95% CI 2-sided [0.96 to 2.05]

ADVERSE EVENTS:
Arm/Group | Varenicline and Buproprion SR | Varenicline and Placebo
Serious Adverse Events (participants affected / at risk) | 6/249 | 6/257
Other Adverse Events (participants affected / at risk) | 165/249 | 161/257
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Varenicline and Buproprion SR (N=249) | Varenicline and Placebo (N=257)
trauma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — sustained trauma during a motor vehicle collision
food poisining (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
diverticulitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
deep vein thrombosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) — new diagnosis
pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
death (Immune system disorders) | 0 (0) | 1 (1) — death due to complications from human immunodeficiency virus 6 months after the study drug was discontinued
attempted suicide (Psychiatric disorders) | 0 (0) | 1 (1) — 9 months after the study drug was discontinued
lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Varenicline and Buproprion SR (N=249) | Varenicline and Placebo (N=257)
sleep disturbance (General disorders) | 100 | 91
nausea (Gastrointestinal disorders) | 55 | 54
constipation (Gastrointestinal disorders) | 26 | 19
headache (Nervous system disorders) | 21 | 22
irritability (General disorders) | 21 | 12
anxiety (General disorders) | 18 | 8
difficulty concentrating (General disorders) | 14 | 10
mood disturbance (General disorders) | 13 | 7
dizziness (General disorders) | 10 | 10
abnormal dreams (General disorders) | 9 | 19
restlessness (General disorders) | 9 | 5
depressive symptoms (Psychiatric disorders) | 9 | 2
fatigue (General disorders) | 7 | 17
dry mouth (General disorders) | 7 | 9
dispepsia (Gastrointestinal disorders) | 5 | 1
flatulance (Gastrointestinal disorders) | 1 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes